CLINICAL TRIAL: NCT06777069
Title: Enhanced Palatal Wound Healing With Leucocyte- and Platelet-Rich Fibrin After Free Gingival Graft Harvesting: A Controlled Prospective Clinical Trial
Brief Title: Effect of Leucocyte- and Platelet-Rich Fibrin on Palatal Wound Healing After Free Gingival Graft Harvesting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Serap Gulsever, Principal Investigator, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMUH-OMFS-SG-01
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Wound Healing
Keywords: free gingival graft, platelet rich fibrin, wound healing
MeSH Terms: interventions — Leukocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leucocyte and platelet rich fibrin (L-PRF) (Experimental): The L-PRF membrane was sutured to the palatal donor sites
  Interventions: Procedure: Leucocyte and platelet rich fibrin membrane application
- Control (No Intervention): The palatal donor sites healed by secondary intention without L-PRF application

INTERVENTIONS:
Procedure: Leucocyte and platelet rich fibrin membrane application — Leukocyte and platelet rich membrane, obtained by centrifuging 10 ml of venous blood collected from the patient's antecubital vein, was sutured to the donor sites.
  Arms: Leucocyte and platelet rich fibrin (L-PRF)

SUMMARY:
Autogenous palatal free gingival graft harvesting presents challenges for patients due to the increased risk of postoperative morbidity related to a second intraoral surgical wound that heals with secondary intention. This study aimed to evaluate the efficacy of the application of leukocyte- and platelet-rich fibrin (L-PRF) membrane to the palatal donor site on wound healing, hemostasis, and pain control after free gingival graft harvesting. Twenty-six adult patients with insufficient attached gingiva underwent soft tissue augmentation using free gingival grafts harvested from the palate. Patients were randomized to either an L-PRF group or a control group. In the L-PRF group, the L-PRF membrane was sutured to the donor sites, whereas in the control group, donor sites healed by secondary intention. Postoperative evaluations were conducted on days 1, 3, 5, and 7 and at weeks 2, 3, 4, 5, and 6. Donor sites were evaluated clinically for pain, burning sensation, bleeding, wound healing, and color match to adjacent tissues. Donor site wound areas were analyzed using digital images.

DETAILED DESCRIPTION:
Soft tissue grafting techniques using autogenous free gingival grafts and connective tissue grafts are reliable and predictable procedures that are commonly used to increase the dimensions of keratinized gingiva. These tehniques are indicated in situations such as shallow vestibular depth, gingival recession, and inadequate peri-implant attached gingiva. Although free soft tissue grafts can be harvested from various intraoral sites, the keratinized gingiva of the hard palate in the premolar-molar region is the most commonly used donor site. However, harvesting tissue from the palate presents challenges for patients, including a second intraoral surgical wound and an increased risk of postoperative morbidity. The palatal wound, which typically heals over two to four weeks by secondary intention, often causes significant patient discomfort due to pain, burning sensation, prolonged bleeding, and delayed healing, often caused by secondary irritation.

Leukocyte- and platelet-rich fibrin (L-PRF), a second-generation platelet concentrate, was developed for oral and maxillofacial surgery in 2001 by Choukroun et al. Polymerization without any biochemical activation, which occurs in a manner comparable to the natural coagulation process, produces a strong fibrin matrix resistant to rapid resorption. Compressing this fibrin matrix creates a strong, suture-resistant membrane that can be fixed to the wound edges and provides a stable barrier against the oral environment.

While L-PRF has shown promise in several applications in regenerative dentistry, randomized controlled clinical trials evaluating L-PRF membrane as an adjunct for donor site wound healing in free gingival grafting procedures are limited in the literature. This study aimed to evaluate the efficacy of L-PRF membrane as a palatal wound dressing in promoting wound healing, hemostasis, and pain control at palatal donor sites following free gingival grafting procedures.

Patients requiring soft tissue augmentation with a free gingival graft due to inadequate keratinized attached gingiva were included in this study. Patients were randomized to either an L-PRF group (n=13) or a control group (n=13). All procedures were performed by a single clinician to reduce variability in surgical technique. After achieving adequate anesthesia, a recipient site was prepared to receive the graft in areas lacking sufficient attached gingiva. This procedure involved an incision at the mucogingival junction followed by blunt dissection to separate the epithelium from the underlying connective tissue, creating a vascular bed for graft integration and survival. A sterile paper template was created to match the dimensions of the recipient site. The paper template was positioned on the palatal mucosa in the premolar/molar region, and the graft margins were outlined with a scalpel. A 1-2 mm thick graft consisting of epithelium and a thin layer of connective tissue was carefully harvested by moving the blade parallel to the mucosal surface. The free gingival graft was carefully oriented on the recipient site, with the epithelium facing outward and the connective tissue in contact with the recipient bed. It was then sutured to ensure close contact between the graft and the underlying tissue to prevent any movement that could compromise revascularization and lead to graft failure. In the L-PRF group, 10 ml of venous blood was drawn from the antecubital vein of the patient using sterile, anticoagulant-free vacutainer tubes and immediately centrifuged at 3000 rpm for 10 minutes. A fibrin clot was structured in the middle of the tube, just between the red corpuscles at the bottom and the acellular plasma at the top. The L-PRF layer was isolated and compressed into a flexible membrane using its special box. The L-PRF membrane was shaped to fit the donor site wound and placed as a single layer, ensuring complete contact with the underlying tissue. It was secured at the wound corners using 5-0 bioabsorbable polyglactin sutures to minimize displacement during the healing process.

Participants were evaluated on days 1, 3, 5, and 7, and weeks 2, 3, 4, 5, and 6 postoperatively to monitor wound healing and complications at the palatal donor site. An examiner recorded subjective parameters (pain, burning sensation), clinically evaluated objective parameters (postoperative bleeding, wound healing, and color matching with the adjacent healthy tissue), obtained donor site photographs, and performed wound area measurements using digital image analysis. Blinding of patients to L-PRF treatment was not feasible due to ethical concerns regarding the collection of blood samples in the control group, and blinding of investigators during digital image analysis and clinical assessment was also not feasible due to the nature of the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

- Patients requiring soft tissue augmentation with a free gingival graft due to inadequate keratinized attached gingiva (shallow vestibular depth, gingival recession)

Exclusion Criteria:

* Patients under 18 years of age
* Patients with systemic medical conditions that may compromise wound healing (e.g., uncontrolled diabetes mellitus, hypertension, blood disorders, rheumatoid arthritis)
* Patients receiving medication that may affect periodontal tissues (e.g., antibiotics, immunomodulatory drugs, steroids, non-steroidal anti-inflammatory drugs) within the last 3 months before surgery
* Patients receiving anticoagulant and antiaggregant therapy
* Smokers
* Pregnancy or breastfeeding
* History of palatal free gingival graft harvesting procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Donor site pain | Postoperative day 1 and weeks 1, 2, 3, and 4
  Pain at the donor site was assessed using a VAS (Visual Analogue Scale) of 0-10.

SECONDARY OUTCOMES:
Donor site burning sensation | Postoperative day 1 and weeks 1, 2, 3, and 4
  Burning sensation at the donor site was assessed using a VAS(Visual Analogue Scale) of 0-10.
Donor site bleeding | Postoperative days 1, 3, 5, and 7
  Postoperative bleeding at the palatal donor site was assessed using a scale of 0 to 3: 0 = no bleeding, 1 = mild bleeding, 2 = moderate bleeding, and 3 = severe bleeding.
Donor site color matching with the adjacent healthy tissue | Postoperative day 1 and weeks 1, 3, and 6
  The color matching of the donor site with the adjacent healthy tissue was assessed using a scale of 0 to 10: 0 = no match, 10 = perfect match.
Donor site clinical healing | Postoperative weeks 1, 2, 3, and 4
  Clinical wound healing at the donor site was scored from 0 to 5 based on the consistency of the clinical appearance with the expected course of healing. Deviations from the expected appearance were recorded as "-1". The expected healing course was as follows: Days 1-7: Fibrin covers the wound surface with petechiae at the wound edge; Days 7-14: Decreased fibrin coverage; Days 14-21: Epithelialization of the defect area; Day 21 onwards: Complete healing.
Donor site wound area | At baseline, on postoperative day 3, and at weeks 1, 2, 3, and 4
  Donor site wound areas were measured digitally from standardized photographs taken using an occlusal mirror.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Gulsever, DDS, PhD, Principal Investigator — Medipol University
Locations (1):
- Baskent University, Faculty of Dentistry, Çankaya/Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We are planning to share our data, after publication of the study
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after application
Access Criteria: via e-mail